CLINICAL TRIAL: NCT03059680
Title: Safety and Physiologic Effects of Implementing a High Potassium Diet in Heart Failure Patients
Brief Title: Effects of Implementing a High Potassium Diet in Heart Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSH 11-0259-A
Record Dates: First submitted 2017-02-16; First posted 2017-02-23 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Heart Failure
Keywords: Potassium; Nutrition
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Masking Description: Treating physicians and participants were not blinded to randomization. Investigators performing randomization and analysis of dietary intake were blinded.
Oversight: Data Monitoring Committee: No

ARMS (2):
- High potassium diet group (Experimental): Individuals in this arm were asked to increase dietary potassium intake over a 4 week period. This was achieved through an increase in consumption of fruits and vegetables.
  Interventions: Other: High potassium diet
- Usual diet group (No Intervention): Individuals in this group were asked to continue habitual dietary intake

INTERVENTIONS:
Other: High potassium diet — An increase in consumption of high potassium fruits and vegetables
  Arms: High potassium diet group

SUMMARY:
This study evaluates the safety and physiologic effects of increasing dietary potassium intake in individuals with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* All patients classified as having HF, both systolic and diastolic.
* New York Heart Association class II-III symptoms.
* Treatment with an beta blocker, ACE inhibitor, or angiotensin receptor blocker without any adjustment over the previous month
* Intake at baseline of ≤ 3 servings of fruits and vegetables per day. Servings defined by Health Canada's food guide.

Exclusion Criteria:

* Patients with an episode of decompensated heart failure, acute coronary syndrome, or revascularization within the previous 3 months of study inclusion.
* Patients receiving insulin therapy
* Glomerular filtration rate < 40mL/min/1.73 m2
* Pregnancy and lactation (women of childbearing potential will be included but will have to have a negative pregnancy test prior to inclusion).
* Inability to provide informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Serum potassium concentration | 10 days and 3 weeks

IPD SHARING:
Plan to Share IPD: No